CLINICAL TRIAL: NCT01765868
Title: A Human Phase I Absolute Bioavailability Study of PRT054021 in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-012
Record Dates: First submitted 2012-12-28; First posted 2013-01-10 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Healthy Subjects
Keywords: Betrixaban; Healthy; Bioavailability
MeSH Terms: interventions — betrixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Oral and IV Betrixaban (Experimental)
  Interventions: Drug: Betrixaban

INTERVENTIONS:
Drug: Betrixaban — Single Oral dose 80 mg betrixaban and Single IV (15 ml) carbon 14 80 micrograms Betrixaban administered over 15 minutes, 2 hours after the oral dose

SUMMARY:
This is a open label, single center, single oral dose, study of PRT054021, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men ages of 19 and 65 years old, inclusive
* BMI of 18-35 kg/m2

Exclusion Criteria:

* Clinically significant comorbid disease
* History of substance abuse

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percent of orally absorbed dose | over 72 hours